CLINICAL TRIAL: NCT00196521
Title: A Clinical Evaluation of the Tension-Free Vaginal Tape Obturator System For Treatment of Stress Urinary Incontinence
Brief Title: A Clinical Evaluation of the Tension-Free Vaginal Tape Obturator System For Treatment of Stress Urinary Incontinence (Urinary Leakage)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ethicon, Inc. (Industry)
Responsible Party: Ethicon, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 300-04-004
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2007-12-13 (Estimated); Status verified 2007-03

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Tension-free vaginal tape obturator system

SUMMARY:
Stress urinary incontinence affects nearly 30 million women worldwide and the main goal of surgical treatment is to stop urinary incontinence (urinary leakage) that occurs with physical activity, coughing, sneezing, etc.Patients in the study will have an operation to improve urinary incontinence symptoms. This will involve inserting a mesh sling to help support the urethra (tube leading into your bladder). During the operation, the study doctor will use tension-free vaginal obturator system. The study will include women diagnosed with Stress Urinary Incontinence who have completed their families.

ELIGIBILITY:
Inclusion Criteria:

* Patient has objective demonstrable signs of stress urinary incontinence (SUI), including patients with ISD. Objective testing includes: standing stress test, urodynamics evaluation, or pad test.
* Patient is age 18 or older.
* Patient had a hysterectomy, tubal ligation or is otherwise incapable of pregnancy, or had a negative pregnancy test prior to study entry and has decided to cease childbearing.
* Patient agrees to participate in the study, including completion of all study-related procedures and evaluations, and documents this agreement by signing the IRB/EC-approved informed consent.

Exclusion Criteria:

* Patient has an associated or suspected neurological disease.
* Patient is on anti-coagulation therapy.
* Patient has received an investigational drug or device in the past 60 days.

For patients having URP measurements at selected sites:

* Patient has an active lesion or present injury to perineum or urethra.Patient has a urethral obstruction.
* Patient has an unreduced cystocele > Stage 1. (Reduction of prolapse prior to URP testing is required.) Reduction of Cystocele (if applicable). Patients should be seated in a semi-fowler's position with head of bed at 40-60 degrees.

Carefully place a half of a speculum into the vagina, reducing prolapse to less than stage 1. Be careful not to over extend or elongate the vaginal length.

The half of a speculum must be placed with pressure emphasis on the posterior and apical areas. Anterior wall pressure or urethral pressure must be avoided at all times.

* The subject has active infection upon urine dipstick analysis, defined as ≥+1 leukocytes or ≥+1 nitrates (Must reschedule appointment after UTI resolves.)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2005-01; Study Completion 2007-03

PRIMARY OUTCOMES:
Overall incidence of treatment success.

SECONDARY OUTCOMES:
Assessment of unresolved de novo urgency post-treatment.
No additional surgery required to correct SUI post-treatment
Intraoperative and postoperative complications
Quality-of-life measurements
Return to usual activity
Patient satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Martin Weisberg, MD, Study Director — Ethicon, Inc.
Locations (19):
- United States (11):
  - Urogynecology Associates of CO, Denver, Colorado
  - Bladder Control Center, Norwalk, Connecticut
  - Urogynecology Specialists of Kenuckiana, Louisville, Kentucky
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Oakwood Hospital, Dearborn, Michigan
  - Sheldon Freedman, MD, Las Vegas, Nevada
  - St. Peter's University Hospital, New Brunswick, New Jersey
  - The Institute for Female Pelvic Medicine & Reconstructive Surgery, Allentown, Pennsylvania
  - University Urology, Knoxville, Tennessee
  - McDonlad Murrmann Women's Clinic, Memphis, Tennessee
  - Sound Urology Ambulatory Surgery Center, Edmonds, Washington
- Sunnybrook & Women's College Health Sciences Center, Toronto, Ontario, Canada
- France (2):
  - Service d'Urologie, Marseille
  - Hopital Des Diaconesses, Paris
- Klinikum der Eberhard-Karls-Universität, Tübingen, Germany
- Women's and Children's Hospital, Singapore, Singapore
- South Korea (2):
  - Samsung Medical Center, Seoul
  - University of Ulsan College of Medicine and Asan Medical Center, Seoul
- Southport District General Hospital, Southport, United Kingdom